CLINICAL TRIAL: NCT01808846
Title: Neural Functioning of Feeding Centers in Obese Youth
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sonia Caprio, Professor of Pediatrics, Yale University
Other Study IDs: 1001006251; R01DK085577 (NIH)
Record Dates: First submitted 2012-10-30; First posted 2013-03-11 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin Resistance; functional magnetic resonance imaging; glucose; fructose; hypothalamus; neuronal circuits; feeding behavior
MeSH Terms: conditions — Obesity; Insulin Resistance; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lean Adolescents: Kids aged 12-17 with body mass index less than 25% and normal glucose tolerance test results
- Obese Insulin Sensitive: Obese Insulin Sensitive Adolescents aged 12-17 with BMI>95th% and whole body insulin sensitivity index > 3.
- Obese Insulin Resistant Adolscent: Obese Insulin Resistant Adolescents 12-17 with BMI> 95th% and WBISI<1.2.

SUMMARY:
To explore whether obese adolescents with insulin resistance and relative low leptin levels exhibit functional alterations of the neuronal circuits involved in the regulation of energy metabolism and food seeking behaviors.

We here propose to test the hypothesis that the reward circuitry is dysregulated in obese adolescents and is related to the degree of insulin resistance and hyperinsulinemia.

DETAILED DESCRIPTION:
Functional Magnetic Resonance Imaging (fMRI) provides a non-invasive method to assess the functional pathways affected by nutrient ingestion and therefore can help answer important questions regarding potential differences in the response of brain regions involved in feeding.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescents
* Good general health,
* taking no medication on a chronic basis
* Age 12 to 17 yrs,
* in puberty (girls and boys: Tanner stage II - IV)

Obese Insulin Resistant Adolescents

* (BMI> 95th)
* (WBISI<1.2 plus a low adiponectin <6 ug/dl and
* high triglyceride levels >130mg/dl)

Obese Insulin Sensitive Adolescents

* (BMI>95th)
* (WBISI >3) plus high adiponectin >8 ug/ml and
* triglyceride levels > 80 mg/dl Girls who begin menstruating must have a negative pregnancy test during the study

Eligibility criteria for healthy non-obese children and adolescents:

* Brother or sister with obesity
* Age 12 to 17 years
* Normal fasting glucose and lipids in the child, and
* normal OGTT
* No use of any medication known to affect glucose, lipid metabolism and inflammation
* No endocrinopathies
* No use of any antipsychotic medication
* BMI >25th to <75th ( Center for Disease Control (CDC) BMI Charts)
* Minimum weight of 90lbs (CDC Growth Charts)

Exclusion Criteria

* Baseline creatinine >1.0 mg
* Pregnancy
* Presence of endocrinopathies (e.g. Cushing syndrome)
* Cardiac or pulmonary or other significant chronic illness
* Adolescents with psychiatric disorder or with substance abuse determined via self-report.
* Use of anorexic agents No metal implants

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Clinic patients of Dr. Caprio at the Yale Pediatric Obesity Clinic who have undergone oral glucose tolerance testing (OGTT) and found to be insulin resistant or sensitive and/or previous research subjects who were found to be insulin resistant or sensitive and who agreed to be contacted for other studies will be contacted.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
measure of cerebral blood flow response to glucose ingestion | Baseline and 2 year follow up
  fmri on 3T to measure blood flow response after ingestion of glucose drink

SECONDARY OUTCOMES:
measure of cerebral blood flow response to fructose ingestion | Baseline and 2 year follow up
  fmri on 3T to measure blood flow response after ingestion of fructose drink

OTHER OUTCOMES:
measure of BOLD signal brain reactivity to food cues | Baseline and 2 year follow up
  fmri on 3T to measure blood flow response to visually presented food cues

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jastreboff AM, Sinha R, Arora J, Giannini C, Kubat J, Malik S, Van Name MA, Santoro N, Savoye M, Duran EJ, Pierpont B, Cline G, Constable RT, Sherwin RS, Caprio S. Altered Brain Response to Drinking Glucose and Fructose in Obese Adolescents. Diabetes. 2016 Jul;65(7):1929-39. doi: 10.2337/db15-1216. Epub 2016 Apr 5. PMID 27207544
- [Derived] Jastreboff AM, Lacadie C, Seo D, Kubat J, Van Name MA, Giannini C, Savoye M, Constable RT, Sherwin RS, Caprio S, Sinha R. Leptin is associated with exaggerated brain reward and emotion responses to food images in adolescent obesity. Diabetes Care. 2014 Nov;37(11):3061-8. doi: 10.2337/dc14-0525. Epub 2014 Aug 19. PMID 25139883